CLINICAL TRIAL: NCT05608759
Title: Effect of a Home-based, Supervised Prehabilitation With Wearable Technology for Patients With Non-small Cell Lung Cancer Before Lung Resection: a Single-arm, Prospective Study
Brief Title: Exercise Prehabilitation for Patients With NSCLC Before Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Zhang Ni, Professor, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TJ-IRB20220564
Record Dates: First submitted 2022-10-27; First posted 2022-11-08 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Prehabilitation; Non Small Cell Lung Cancer; Cardiorespiratory Fitness; Surgery
Keywords: Prehabilitation; Cardiorespiratory fitness; Non-small cell lung cancer; Exercise; Wearable technology; Surgery
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): 4 weeks of multimodal pre-rehabilitation
  Interventions: Behavioral: Multimodal prehabilitation

INTERVENTIONS:
Behavioral: Multimodal prehabilitation — 4 weeks of an supervised, pre-operative exercise prescription augmented by a wearable fitness device.

SUMMARY:
To explore the safety and compliance of a wearable telemedicine device that can receive basic vital signs in real time, and its active supervision mode with real-time adjustment of exercise prescription for preoperative prehabilitation exercises in patients at home; and to evaluate the effectiveness of preoperative prehabilitation exercises in a telemedicine active supervision mode in patients undergoing thoracoscopic lung tumour resection, taking into account the patient's cardiopulmonary exercise test, postoperative complications and quality of life scores.

ELIGIBILITY:
Inclusion Criteria:

1. Capacity to give informed consent.
2. Are able to tolerate surgery (i.e., segmentectomy, lobectomy) as indicated by standard clinical pre-op evaluation, including pulmonary function tests and cardiopulmonary exercise testing.
3. Patients who can use a smartphone application.
4. Patients who are diagnosed of stage I or II Non-small-cell lung carcinoma (NSCLC) diagnosis, with or without pre-operative histologic confirmation.
5. Patients who can perform an exercise program for at least 4 weeks from the first visit to the preoperative clinic to elective surgery.

Exclusion Criteria:

1. Known contraindication for cardiopulmonary exercise testing.
2. Patients who have a major medical or psychiatric disorder that is expected to affect exercise.
3. Pregnancy or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity | Baseline, 4 weeks after prehabilitation exercise
  Exercise testing on a cycloergometer(VO2 max)

SECONDARY OUTCOMES:
Forced expiratory volume in 1 s(FEV1) | Baseline, 4 weeks after prehabilitation exercise, 7 days after surgery, 30 days after surgery
  Forced expiratory volume in 1 s (FEV1) of pulmonary function will be measured in liters
Forced vital capacity (FVC) | Baseline, 4 weeks after prehabilitation exercise, 7 days after surgery, 30 days after surgery
  Forced vital capacity (FVC) of pulmonary function will be measured in liters.
Acceptance of technology | 4 weeks of prehabilitation exercise
  number of hours the fitness tracker was worn in pre-operative period
Change in quality of life | Baseline, 4 weeks after prehabilitation exercise, 7 days after surgery, 30 days after surgery
  as assessed by the EORTC QLQ C30 questionnaire
Change in grip-strength | Baseline, 4 weeks after prehabilitation exercise, 7 days after surgery, 30 days after surgery
  Grip strength per dynamometer
Length of stay in hospital | Up to 30 postoperative days
  Number of days from surgery to discharge home
Post-operative complications | From day of surgery to 30-days afterwards
  Classified using the Clavien Dindo Classification
Adherence to exercise | 4 weeks of prehabilitation exercise
  number of completed pre-operative exercise sessions divided by number of prescribed sessions, according to exercise log

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

REFERENCES:
- [Derived] Sun Q, Omindo WW, Liu W, Huang Y, Zhang R, Qian Y, Li X, Qiu R, Zheng S, Ping W, Zhang N. Your preoperative rehabilitation assistant: A study protocol for the impact of a telemedicine-supported preoperative home rehabilitation program on the prognosis of patients undergoing thoracoscopic surgery. Digit Health. 2024 Jun 5;10:20552076241258362. doi: 10.1177/20552076241258362. eCollection 2024 Jan-Dec. PMID 39351312